CLINICAL TRIAL: NCT05332366
Title: A Phase 2a, Randomized, Double-Blind, Vehicle-Controlled, Single Site, Exploratory Trial to Assess the Effect of Delgocitinib Cream 20 mg/g on the Molecular Signature, Safety, and Efficacy in Adults With Frontal Fibrosing Alopecia
Brief Title: A Trial to Assess the Effect of Delgocitinib Cream 20 mg/g on the Molecular Signature, Safety, and Efficacy in Adults With Frontal Fibrosing Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXP-2228
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Frontal Fibrosing Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Delgocitinib - Delgocitinib (Experimental): Participants were blinded and randomised to delgocitinib cream treatment for the first 12 weeks, followed by an open label treatment with delgocitinib cream treatment for another 12 weeks.
  Interventions: Drug: Delgocitinib cream
- Placebo - Delgocitinib (Placebo Comparator): Participants were blinded and randomised to placebo cream treatment for the first 12 weeks, followed by an open label treatment with delgocitinib cream treatment for another 12 weeks.
  Interventions: Drug: Delgocitinib cream; Drug: Delgocitinib cream vehicle
- No treatment (No Intervention): Participants did not receive any treatment. They only provided a molecular signature of healthy skin to act as a control.

INTERVENTIONS:
Drug: Delgocitinib cream — Cream for topical application
  Other Names: LEO 124249 cream
  Arms: Delgocitinib - Delgocitinib; Placebo - Delgocitinib
Drug: Delgocitinib cream vehicle — The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
  Arms: Placebo - Delgocitinib

SUMMARY:
This purpose of this trial was to investigate the molecular signature of frontal fibrosing alopecia (FFA) and the effect of delgocitinib cream 2% on reversing the FFA disease signature in active lesions. The trial also investigated the clinical effect of delgocitinib cream on FFA compared to a placebo cream.

ELIGIBILITY:
Inclusion criteria

For Group 1 only (subjects with FFA):

1. Male or female subject aged 18 years of age or older at the time of consent.
2. Subject has clinically confirmed diagnosis of FFA.
3. Subject has a target area with a perifollicular erythema score ≥ 2 and a perifollicular scale score ≥ 2 at Screening and Day 1.

For Group 2 only (healthy subjects):

1. Female subject aged 45 years of age or older at the time of consent.
2. Female is postmenopausal.
3. Subject is in good general health.

Exclusion criteria

For all subjects:

1. Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the trial.
2. Presence of hepatitis B or C infection or HIV infection at screening.

For Group 1 only (subjects with FFA):

1. History of other scalp/hair disease including discoid lupus erythematosus and central centrifugal cicatricial alopecia.
2. Subject who has undergone scalp reduction surgery or hair transplantation.
3. Subject is known to have immune deficiency or is immunocompromised.
4. Subject has used intralesional scalp corticosteroids or platelet rich plasma injection in the last 4 weeks prior to randomization.
5. Subject has used systemic treatment with immunosuppressive/modulating medication or medication within 4 weeks prior to randomization.
6. Subject has used any topical medicated treatment that could affect FFA within 2 weeks prior to randomization.
7. Subject has received any phototherapy within 4 weeks prior to randomization.

For Group 2 only (healthy subjects):

1. Subject has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the trial assessments.
2. Subject has used a topical medicated treatment on the targeted skin sites within 2 weeks prior to trial assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Translational Medical Leader, Study Director — LEO Pharma
Locations (1):
- LEO Investigational Site, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin A, Shokrian N, Kelley KJ, Correa da Rosa J, Del-Duca E, Bissonnette R, Sorensen OE, Nielsen AB, Guttman-Yassky E, Senna MM. Randomized Controlled Trial of the Topical Jak Inhibitor Delgocitinib Cream in Patients with Frontal Fibrosing Alopecia. J Invest Dermatol. 2025 Oct 14:S0022-202X(25)03406-2. doi: 10.1016/j.jid.2025.09.375. Online ahead of print. PMID 41101628

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in the United States and consisted of 2 cohorts: Cohort 1 included 30 subjects with FFA and Cohort 2 included 5 healthy postmenopausal female subjects. Both cohorts were conducted in parallel.
Pre-assignment Details: Eligible subjects were randomized into the trial after a screening period. They were assigned to receive either delgocitinib cream or a placebo twice daily for 12 weeks. After completing this period, they continued using delgocitinib cream for another 12 weeks.
Period: Overall Study
Arm/Group | Delgocitinib - Delgocitinib | Placebo - Delgocitinib | No Treatment
Started | 15 | 15 | 5
Completed | 15 | 15 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Treatment: Participants did not receive any treatment. They will only provide a molecular signature of healthy skin to act as a control.
- Total: Total of all reporting groups
Arm/Group | Delgocitinib - Delgocitinib | Placebo - Delgocitinib | No Treatment | Total
Number analyzed (Participants) | 15 | 15 | 5 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (6.82) | 62.6 (12.64) | 67.4 (9.81) | 64.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 5 | 35
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 13 | 15 | 5 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 15 | 5 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 5 | 35
Height (cm) [Mean (Standard Deviation); unit: units on a scale] | 163.34 (7.557) | 162.49 (6.970) | 165.20 (8.415) | 163.24 (7.257)
Weight (kg) [Mean (Standard Deviation); unit: units on a scale] | 68.41 (15.245) | 75.41 (16.503) | 72.40 (17.418) | 71.98 (15.950)

OUTCOME MEASURES:

1. Primary Outcome: Change in Expression of Chemokine (C-X-C Motif) Ligand 9 (CXCL9), Chemokine (C-X-C Motif) Ligand 10 (CXCL10), and Interferon (IFN)-γ From Baseline to Week 12.
Description: CXCL9, CXCL10 and IFN-γ are small proteins that act as chemical messengers, especially in the immune system.
Time Frame: Baseline and Week 12
Population: No data was collected for "No Treatment" Arm/Groups".
Measure: Number; unit: Fold-changes
Arm/Group | Delgocitinib - Delgocitinib | Placebo - Delgocitinib | No Treatment
Number analyzed (Participants) | 15 | 15 | 0
Fold-changes
  (C-X-C motif) ligand 9 (CXCL9) | -3.10 | -1.12 |
  Chemokine (C-X-C motif) ligand 10 (CXCL10) | -2.60 | -1.10 |
  Interferon (IFN)-γ | -1.49 | -1.097 |

2. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) From Baseline to Week 12.
Description: Treatment emergent adverse events (TEAEs) were defined as any AEs with onset date on or after the first study treatment dosing.
Time Frame: Between baseline and Week 12
Population: No investigational product was administered in Cohort 2 "No Treatment" Arm/Groups" and thereby were no treatment-emergent AESIs reported in this trial for "No Treatment" Arm/Groups".
Measure: Number; unit: events
Arm/Group | Delgocitinib - Delgocitinib | Placebo - Delgocitinib | No Treatment
Number analyzed (Participants) | 15 | 15 | 0
events | 4 | 9 |

ADVERSE EVENTS:
Time Frame: Baseline and week 12
Description: No investigational product was administered for 'No Treatment' Arm/Groups; and thus collection of adverse events did not occur for the participants in this group.
Groups:
- Placebo - Delgocitinib: Participants were blinded and randomised to placebo cream treatment for the first 12 weeks, followed by an open label treatment with delgocitinib cream treatment for another 12 weeks.
  Delgocitinib cream: Cream for topical application Delgocitinib cream vehicle: The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
Arm/Group | Delgocitinib - Delgocitinib | Placebo - Delgocitinib | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/0
Other Adverse Events (participants affected / at risk) | 6/15 | 10/15 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib - Delgocitinib (N=15) | Placebo - Delgocitinib (N=15) | No Treatment (N=0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 7 (7) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site rash (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Antinuclear antibody positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT05332366/Prot_SAP_000.pdf